CLINICAL TRIAL: NCT03887585
Title: Modified Percutaneous Achilles Tendon Lengthening by Triple Hemisection for Achilles Tendon Contracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, vice dean, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tendon
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Achilles Tendon Contracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Achilles tendon lengthening (Experimental): Surgery of percutaneous Achilles tendon lengthening by triple hemisection
  Interventions: Procedure: Achilles tendon lengthening

INTERVENTIONS:
Procedure: Achilles tendon lengthening — Achilles tendon lengthening by triple hemisection for Achilles tendon contracture

SUMMARY:
This study aims to evaluate the efficacy and safety of this new therapeutic method, which is based on the percutaneous sliding technique with three hemi-cuts in the tendon.

DETAILED DESCRIPTION:
This study aims to provide a new therapeutic theory which bases on the percutaneous sliding technique with three hemi-cuts in the tendon. In this study, Achilles tendon parenchymal at distal level is hemisected through the most distal incision, Achilles tendon parenchymal at proximal level is hemisected through the middle incision, then Achilles tendon lengthening is accomplished by the sliding tendon under forceful dorsiflexion. It can better achieve soft tissue balance and reduce the recurrence of Achilles tendon contracture when Achilles tendon strength in plantarflexion is weakened. Thus in this study, the partial aponeurosis of gastrocnemius is cut off at most proximal incision in order to weaken Achilles tendon strength in plantarflexion.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than three years old;
* Severe Achilles tendon contracture and equinus;
* The time after Achilles tendon contracture more than 6 months ;
* Initial Achilles tendon lengthening.

Exclusion Criteria:

* Patients younger than 3 years;
* The course of Achilles tendon contracture is within 6 months;
* Patients who have suffered from the Achilles tendon lengthening;
* Obvious contracture of other soft tissues occurs in combination, such as compartment syndrome or extensive scar tissues in calf;
* Osteotomy or tendon transposition is needed.
* Ankle joint is damaged obviously, such as Charcot's joint or Hemophilic arthritis;
* Skin soft-tissue infection in the lower limb.
* Initial Achilles tendon lengthening.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the American Orthopaedic Foot & Ankle Society (AOFAS) scores | Before surgery and up to 8 years after surgery
  The AOFAS scores of the patients before and after surgery are recorded. The scale ranges from 0-100 points, and increases of the value represent a better outcome.

SECONDARY OUTCOMES:
Equinus recurrence rate | Up to 8 years after surgery
  The equinus recurrence rate of the patients after surgery is recorded. Lower value represents a better outcome.
Infection rate | Up to 8 years after surgery
  The infection rate of the patients after surgery is recorded. Lower value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Duan, MD, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, China